CLINICAL TRIAL: NCT03328143
Title: Feasibility of Aromatherapy in an Awake Craniotomy Environment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17.101
Record Dates: First submitted 2017-10-27; First posted 2017-11-01 (Actual); Results first posted 2024-08-05 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-07

CONDITIONS: Intracranial Pathology
Keywords: Craniotomy, anxiety, malignant, cancer, brain tumor
MeSH Terms: conditions — Anxiety Disorders; Neoplasms; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment with Lavender (Experimental): Lavender (Lavandula angustifolia) aromatherapy will be administered at regular intervals using a nasal inhaler.
  Interventions: Drug: Lavender (Lavandula angustifolia)

INTERVENTIONS:
Drug: Lavender (Lavandula angustifolia) — Lavender (Lavandula angustifolia) is an essential oil.

SUMMARY:
Awake craniotomy for tumor surgery allows for mapping of speech, motor and sensory function during tumor resection. Awake craniotomy is increasingly utilized as it has several advantages over a traditional general anesthetic technique. Though many patients tolerate awake cranial surgery well, recent studies found that roughly 30% of patients experience moderate to severe pain and anxiety, while 50% report moderate fear and 11% report severe fear. Therefore, alternative methods to mitigate pain, anxiety, and fear are needed. In this study, the investigators will employ lavender aromatherapy to reduce anxiety and improve the satisfaction with pain control.

DETAILED DESCRIPTION:
The lavender aromatherapy trial protocol was developed in conjunction with the Aurora Health Care (AHC) Integrative Medicine Department and Certified Clinical Aromatherapy Practitioners (CCAP). Participating patients received standard of care intraoperative analgesic and anxiolytic management plus lavender aromatherapy. Lavender scent was administered via nasal inhaler. The lavender essential oil, base oil, and nasal inhaler were provided by AHC Integrative Medicine Department to ensure standardization across all patients. The nasal inhaler was prepared with 15 gtts (drops) of lavender essential oil and 4 gtts (drops) of the base oil (grapeseed oil). A CCAP from Integrative Medicine provided training on the delivery of lavender aromatherapy to all study team members. This person consulted on the participation of the first three subjects and was present in the operating room (OR) to oversee administration of lavender aromatherapy. The CCAP was also available for consultation during the course of the study, as needed.

A dedicated OR nurse, neuropsychologist, or neuropsychometrist oversaw administration of lavender aromatherapy to subjects. They monitored the subject during study participation and were prepared to discontinue the trial if they felt continued participation was detrimental to the patient. Lavender aromatherapy was administered for up to five minutes using the nasal inhaler at designated time points (preoperative, induction) and every 30 minutes during the surgery. Although the majority of the time OR personnel administered the aromatherapy, some patients were able to and chose to self-administer. Additional lavender aromatherapy treatments were provided at any time upon request. During non-use periods, the nasal inhaler was capped and sealed. If the subject was unable to verbally request the research team member to hold the nasal inhaler under their nose, the subject's participation in the study was terminated. Additionally, subjects were free to discontinue administration of aromatherapy at any time during their participation in the study. The timing and reason of discontinuation of lavender aromatherapy was recorded.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient aged 18 and older undergoing awake cranial neurosurgery

Exclusion Criteria:

* Allergy or sensitivity to the aromatherapy agent (Lavender)
* Aversion to lavender scent
* History of asthma, chronic obstructive pulmonary disease (COPD)
* History of contact dermatitis following exposure to cosmetic fragrances
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Rovin, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Aurora Health Care, Aurora St. Luke's Medical Center, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 40 patients were enrolled, 31 completed the trial
Groups:
- Lavender Group: Lavender (Lavandula angustifolia) aromatherapy will be administered at regular intervals, or upon request, using a nasal inhaler.
Period: Overall Study
Arm/Group | Lavender Group
Started | 40
Completed | 31
Not Completed | 9
Not completed — Declined | 3
Not completed — Required increased sedation | 4
Not completed — Couldn't smell the lavender in the OR | 1
Not completed — Surgery cancelled | 1

BASELINE CHARACTERISTICS:
Population: The population analyzed are the 31 patients who completed the protocol. All 31 patients received lavender aromatherapy
Arm/Group | Treatment With Lavender
Number analyzed (Participants) | 40
Age, Continuous [Mean (Full Range); unit: years] | 60 [22 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Consented Patients
Description: Determine the number of eligible patients enrolled and consented
Time Frame: From recruitment to end of enrollment period
Measure: Count of Participants; unit: Participants
Arm/Group | Lavender Group
Number analyzed (Participants) | 40
Participants | 40

2. Primary Outcome: Protocol Completion
Description: Determine the number of consented patients completing the trial protocol
Time Frame: From the preoperative evaluation through the post operative evaluation in the Neurosurgical Intensive Care Unit (NICU)
Measure: Count of Participants; unit: Participants
Arm/Group | Lavender Group
Number analyzed (Participants) | 40
Participants | 31

3. Secondary Outcome: Validation of Visual Analogue Scale for Anxiety (VAS-A)
Description: Measure of anxiety, Total Score (0-10). Zero is lowest anxiety, 10 is highest.
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lavender Group
Number analyzed (Participants) | 31
score on a scale | 3.1 (2.968)

4. Secondary Outcome: Validation of Visual Analogue Scale for Pain (VAS-P)
Description: Measure of pain, Total Score (0-10). Zero is lowest level of pain, 10 thee highest
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lavender Group
Number analyzed (Participants) | 31
score on a scale | 1.1 (2.498)

5. Secondary Outcome: Number of Participants Satisfied and Very Satisfied With Pain Treatment Overall.
Description: This is a 5 point Likert scale for the question, "How satisfied are you with your pain treatment overall?" The responses are very dissatisfied, dissatisfied, uncertain, satisfied, very satisfied. The responses are summarized in the data table: Number of Participants Very Dissatisfied with Pain Treatment Overall, Number of Participants Dissatisfied with Pain Treatment Overall, Number of Participants Uncertain About Pain Treatment Overall, Number of Participants Satisfied with Pain Treatment Overall, Number of Participants Very Satisfied with Pain Treatment Overall. A single participant can provide only one response to the question so that the outcome measure Number of Participants Very Dissatisfied with Pain Treatment Overall, for example, means the number of participants very dissatisfied with pain treatment overall. There are not multiple assessments, there are 5 possible responses to the question and, again, only one response is permitted for one patient.
Time Frame: 8 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Lavender Group
Number analyzed (Participants) | 31
Participants
  Very Dissatisfied | 0
  Dissatisfied | 1
  Uncertain | 5
  Satisfied | 12
  Very Satisfied | 13

ADVERSE EVENTS:
Time Frame: From initiation of surgery until discharge from NICU
Arm/Group | Lavender Group
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT03328143/Prot_SAP_000.pdf